CLINICAL TRIAL: NCT04676516
Title: A Phase II Randomized Window of Opportunity Trial Evaluating Clinical and Biological Effects of PRMT5 Inhibitor, GSK3326595, in Early Stage Breast Cancer
Brief Title: A Phase II Window of Opportunity Trial of PRMT5 Inhibitor, GSK3326595, in Early Stage Breast Cancer
Acronym: OTT-19-06
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Ontario Institute for Cancer Research (Other); GlaxoSmithKline (Industry); London Regional Cancer Program, Canada (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OTT-19-06
Record Dates: First submitted 2020-07-28; First posted 2020-12-21 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
Keywords: Window of Opportunity; PRMT5 inhibitor; GSK3326595; Early Stage Breast Cancer; Hormone Receptor (HR) positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — GSK-3326595

STUDY DESIGN:
Intervention Model Description: Phase II, randomized, open label, multi-center, parallel design, window of opportunity trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Participants randomized to treatment with GSK3326595 will be requested to take 15 +/- 3 days of the medication at the dose of 200 mg orally daily (2 capsules of 100 mg) prior to their breast cancer surgery or repeat biopsy. GSK3326595 is a first-in-class small molecule PRMT5 inhibitor in form of an oral capsule.
  Interventions: Drug: GSK3326595
- No Intervention Arm (No Intervention): Participants will receive no treatment for 15 +/- 3 days prior to breast surgery. There is no placebo in this trial.

INTERVENTIONS:
Drug: GSK3326595 — GSK3326595 is a first-in-class small molecule PRMT5 inhibitor in form of an oral capsule.
  Other Names: PRMT5 inhibitor
  Arms: Experimental Arm

SUMMARY:
This is a Phase II Randomized Window of Opportunity Trial Evaluating Clinical and Biological effects of PRMT5 inhibitor, GSK3326595, in Early Stage Breast Cancer

DETAILED DESCRIPTION:
This is a phase II, randomized, open label, multi-center, parallel design, window of opportunity trial in up to 60 patients with early stage Hormone Receptor (HR) positive breast cancer evaluating GSK3326595. In a 2:1 randomization, patients will receive GSK3326595:no treatment for 15 +/- 3 days prior to breast surgery. There is no placebo in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with newly diagnosed histologically confirmed primary invasive breast cancer currently not undergoing any treatment while awaiting surgery
2. Operable breast cancer as assessed by treating surgical oncologist
3. Tumor ≥ 1.0 cm by palpation or imaging
4. ER or PR positive (≥1%) breast adenocarcinoma
5. Her2 negative as per ASCO 2018 guidelines 61
6. Invasive ductal or lobular carcinoma, invasive carcinoma Not Otherwise Specified (NOS)
7. ECOG PS 0-2 (Appendix A)
8. Post-menopausal and not of child bearing potential as defined as: by having 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40mlU/ml and estradiol < 20 pg/mL or have had documented surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks prior.
9. Able to provide written informed consent for the study.
10. Able to swallow and retain orally administered medication.

Exclusion Criteria:

1. Locally Advanced or metastatic breast cancer
2. Prior therapy with chemotherapy or planned neoadjuvant chemotherapy
3. Prior hormonal therapy including tamoxifen, aromatase inhibitors
4. Pre-dominant histology other than invasive ductal or lobular carcinoma
5. Concomitant other invasive malignancy.
6. Hgb < 100 g/L, Platelets < 100 x 10^9 per liter, Absolute Neutrophil Count < 1.5 x 10^9/L
7. Bilirubin ≥ 1.5 times Upper Limit Normal (ULN)
8. ALT ≥ 2.5 times ULN
9. Albumin < 25 g/L
10. INR/PTT > 1.5 times ULN
11. Creatinine clearance calculated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation of less than 50 mL/min/1.73m2.
12. Cardiac abnormalities as evidenced by any of the following:

    1. Baseline QTcF interval ≥ 480 msec
    2. Clinically significant conduction abnormalities or arrhythmias
    3. Presence of cardiac pacemaker or defibrillator with a paced ventricular rhythm limiting ECG analysis.
    4. History or evidence of current ≥ Class II congestive heart failure as defined by New York Heart Association (NYHA).
    5. History of acute coronary syndromes (including unstable angina and myocardial infarction), coronary angioplasty, or stenting within the past 3 months.
    6. Clinically significant cardiomegaly, ventricular hypertrophy, or cardiomyopathy.
13. Any serious known immediate or delayed hypersensitivity reaction(s) to GSK3326595, or idiosyncrasy to drugs chemically related to the investigational drugs.
14. Current use of a prohibited medication or planned use of any forbidden medications during treatment with GSK3326595, which include chemotherapy, immunotherapy, biologic therapy, investigational therapy, or hormonal therapy (other than corticosteroids) while on treatment in this study. GSK3326595 should not be co-administered with potent inhibitors of either BCRP or Pgp such inhibitors include cyclosporine, tacrolimus, and ketoconazole
15. Any clinically significant gastrointestinal (GI) abnormalities that may alter absorption, such as malabsorption syndrome, chronic gastrointestinal disease, or major resection of the stomach and/or bowels that could preclude adequate absorption of the study medication.
16. Severe, uncontrolled systemic disease (respiratory, cardiac, renal, hepatic, bleeding)
17. Currently active liver or biliary disease
18. History of active HIV, Hepatitis B or C infection.
19. Any other criteria which, in the investigator's opinion, renders the patient ineligible to be on study.
20. Subjects with signs/symptoms suggestive of COVID-19 or known COVID-19 positive contacts in the past 14 days would be tested as per local Public Health and/or Institutional Guidelines. If patients are COVID-19 positive at the time of screening, they would be excluded from the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female post-menopausal participants
Enrollment: 40 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Complete cell cycle arrest (CCCA) | 2 years
  The primary outcome is the proportion of patients who achieve a Complete Cell Cycle Arrest (CCCA), defined as a reduction in the proportion of Ki67 positively staining cells to ≤ 2.7%.

SECONDARY OUTCOMES:
Rate of complete cell cycle arrest (CCCA) in patients with wild-type TP53 | 2 years
  The secondary outcome is to assess whether PRMT5 inhibition preferentially results in CCCA in patients with wild-type TP53.
Assess whether PRMT5 inhibition results in reduced expression of ER-α signaling compared to patients with no treatment based on gene expression analysis. | 2 years
  A secondary outcome is to assess whether PRMT5 inhibition results in reduced expression of ER-α signaling.
Assess whether PRMT5 inhibition results in changes in breast-cancer stem cell signature particularly FOXP1 compared to patients with no treatment based on gene expression analysis | 2 years
  A secondary outcome is to assess whether PRMT5 inhibition results in changes in breast-cancer stem cell signature particularly FOXP1.
Perform molecular analysis to identify immunomodulatory effects of GSK3326595 determined by abundance of different immune cells in tumor (CD4, CD8, NK cells, macrophages, etc) in the tumors treated with GSK3326595 alone versus the untreated tumours. | 2 years
  A secondary outcome is to identify the immunomodulatory effects of GSK3326595, by performing exploratory analyses.

OTHER OUTCOMES:
Rate of alternative splicing of Murine Double Minute 4 (MDM4) | 2 years
  A tertiary outcome is to assess if PRMT5 inhibition results in alternative splicing of MDM4.
% of response in participants with high Programmed Cell Death 4 (PDCD4) expression and Cyclin Dependent Kinase Inhibitor 2A (CDKN2A) loss | 2 years
  A tertiary outcome is to assess whether PRMT5 inhibition results in preferential response in patients with high PDCD4 expression and CDKN2A loss.
% of response in participants with defects in homologous recombination DNA repair | 2 years
  A tertiary outcome is to assess whether PRMT5 inhibition results in preferential response in patients with defects in homologous recombination DNA repair.
% of response in participants with defects in Cyclin D (CCND)/ Cyclin-dependent kinases (CDK) pathway | 2 years
  A tertiary outcome is to assess whether PRMT5 inhibition results in preferential response in patients with defects in CCND/CDK pathway.
% of response in patients with defects in phosphatidylinositol-3-kinase (PI3K)/Serine-threonine protein kinase 1 (AKT) pathway | 2 years
  A tertiary outcome is to assess whether PRMT5 inhibition results in preferential response in patients with defects in PI3K/AKT pathway.

CONTACTS AND LOCATIONS:
Overall Officials: John F. Hilton, MD, Principal Investigator — The Ottawa Hospital Cancer Centre
Locations (1):
- St. Joseph's Health Care London, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Researchers may contact Dr. John Hilton for specific requests.